CLINICAL TRIAL: NCT04321915
Title: Study of the Link Between Intestinal Dysbiosis and the Integrity of the Blood Brain Barrier in Autism
Brief Title: Intestinal Dysbiosis and BBB Integrity in Autism
Acronym: LEDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); LBPC, Inserm 1183, IRMB CHU Montpellier (Unknown); UMR 5203, InsermU1191, IGF, Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL18_0197
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: intestinal microbiota; neuroinflammation; brain blood barrier; autism spectrum disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Autism spectrum disorder (Other): Patients will realised quesstionnaires, a blood sample will be collected, the feces will be collected too.
  The analysis of intestinal microbiota and neuroinflammation markers will be processed.
  Interventions: Other: Analysis of intestinal microbiota in autism spectrum desorder; Other: Analysis of neuroinflammation markers in autism spectrum desorder

INTERVENTIONS:
Other: Analysis of intestinal microbiota in autism spectrum desorder — This analysis permit to describe the diversity and composition of microbiota and the factors that may influence them. In fact, the gut microbiota plays a key role in regulating the gut-brain axis
Other: Analysis of neuroinflammation markers in autism spectrum desorder — This analysis permit to reveal the integrity of the blood-brain barrier (BBB) which is affected in autism spectrum desorder.

SUMMARY:
Autism Spectrum Disorder (ASD) is characterised by an impairment of social interactions and communication, associated with repetitive behaviour and restrictive interests. Clinical phenotypes of this neurodevelopmental disorder are heterogeneous and surprisingly up to 70% of ASD patients have gastro-intestinal (GI) disorders, associated with ASD severity and influence by feeding disorders.

Gut-brain axis seems to play a key role in neurodevelopment and ASD pathophysiology. Indeed an intestinal dysbiosis is observed in ASD, as well as intestinal inflammation and permeability. Aspecific inflammatory pattern suggests neuroinflammation processes in ASD. Neuroinflammation is involved in blood brain barrier (BBB) integrity and there are some arguments for a putative BBBimpairment in ASD. Nevertheless, no study has explored all together these parameters in ASD patients.

Here we hypothesise that intestinal dysbiosis in ASD could lead to a BBB impairment through neuroinflammation processes. Furthermore, this association between intestinal dysbiosis and BBB impairment could be influenced by a lot of clinical characteristics, such as ASD severity or GI disorders presence.

The principal aim of our study is to determine if the gut microbiota composition is associated with the BBB integrity in ASD. The secondary objectives are i) too identify in children with ASD some physiopathological pathways involved in this association, with a focus on associations betweenintestinal dysbiosis, intestinal permeability, intestinal permeability, the Th1/Th2 immune response, neuroinflammation and the BBB integrity; ii) to evaluate the influence of these associations on several clinical features of ASD such as ASD severity or GI disorders intensity; iii) to evaluate the influence of nutritional status on biological and clinical parameters.

This study will assess a lot of clinical and biological parameters together, some of them were never explored in ASD children. It will allow to better understand ASD pathophysiology, to highlight new therapeutic pathway, and to promote personalised medicine.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by impaired social interactions and communication, associated with repetitive behaviors and restricted interests. The pathophysiology of ASD is complex due to clinical heterogeneity and numerous comorbidities. Surprisingly, up to 70% of children with ASD have gastrointestinal (GI) disorders, correlated with the severity of ASD. These GI disorders are influenced by eating disorders linked to ASD. There is also an imbalance of the intestinal microbiota in ASD. In addition, the gut microbiota plays a key role in regulating the gut-brain axis. It is involved in brain development and neuroinflammation, one of the pathophysiological tracks in ASD. Neuroinflammation is also involved in regulating the integrity of the blood-brain barrier (BBB), which is affected in ASD. The question if intestinal dysbiosis influences the BBB integrity in ASD therefore arises.

The main objective is to determine if there is an association between the composition of the intestinal microbiota and the integrity of the BBB in ASD.

Secondary objectives are i/ to identify the pathophysiological pathways involved in this association, in particular via the neuroinflammation processes, ii/ to estimate the influence of this association on some ASD characteristics, iii/ to determine the influence of nutritional status on the measured biological and clinical parameters.

This is a monocentric, observational and cross-sectional study of 72 children with ASD, aged 6 to 16, living in the Languedoc-Roussillon region and from the ELENA cohort (this cohort includes 900 French children with an ASD, initially aged 2 to 16, and followed for 6 years).

Serum immunoassays will be assessed for the measurement of neuroinflammation, plasma assays for the intestinal inflammation and permeability. Clinical characteristics will be collected by a clinician and parental questionnaires (ASD severity test, level of social interaction, repetitive and stereotypical behavior, behavioral disorders, quality of life, intensity of GI disorders). Nutritional status will be assessed by serum metabolome analysis and anthropomorphic measures.

Participants will be stratified according to the intensity of their ASD characteristics and the presence or absence of GI disorders.

Descriptive analyses of microbiota composition, biological markers of intestinal permeability and inflammation, neuroinflammation and BBB integrity will be performed using an Heat Map Correlation. Principal component analysis will allow to identify patterns of microbiota compositions. Associations between the different groups of measured biomarkers (microbiota patterns, BBB integrity, intestinal permeability, intestinal inflammation and neuroinflammation) will be performed using multivariate regression models. The models will be systematically adjusted for age and gender.

The study will last 4 and a half years and will end in February 2025. The inclusions will last 42 months. No specific follow-up is planned outside the 6-month maximum period between the study proposal and the inclusion visit. The study will be presented to patients at the end of their visit at 3 or 6 years of follow-up as part of the ELENA cohort. For patients meeting the inclusion criteria and who agrees to participate in the study, two visits will occur at the Center of Autism Ressources of Languedoc-Roussillon (CRA-LR), for the collection of consent and the delivery of the material to be used at home. In the week preceding their second visit to CRA-LR, parents will collect a sample of their child's stool in a dedicated jar which will be packed in a plastic bag and kept in the home-deep-freeze until they reach CRA-LR. A Bristol scale - allowing the display of the child's stools -, a PedsQL GSS questionnaire - evaluating gastrointestinal disorders - and a RBS-R questionnaire - evaluating repetitive and stereotypical behaviors - will be completed by parents. During the inclusion visit, a clinical examination of children will be performed and a blood sample will be collected.

This study will concomitantly assess many clinical and biological parameters, some of whom never explored before in children with ASD. It will allow a better understanding of the implication of the gut-brain axis in the ASD pathophysiology and will open the way to new therapeutic targets.

ELIGIBILITY:
Inclusion criteria:

* Child from the ELENA cohort who received at least 3 years of follow-up in this cohort and a diagnosis of ASD
* Aged 6 to 16 years
* Living in Languedoc-Roussillon
* Consent to participate in the study signed by the legal representative

Exclusion criteria:

* Syndromic autism (neuroanatomical abnormality detected on brain MRI, severe neurological syndrome or polymalformative)
* Known severe gastrointestinal pathology (such as celiac disease or Crohn's disease)
* Other known severe chronic disease (e.g., diabetes)
* Specific diet (gluten-free, casein-free, ketogenic, protein-enriched) within 6 months
* Antibiotics taken within 2 months prior to inclusion
* Probiotics taken in the 6 months prior to inclusion
* Oxytocin intake in the 6 months prior to inclusion
* ADOS Level Module 4 (due to the impossibility of calculating a ADOS-CSS score in this case)
* Not affiliated to a French social security scheme or not beneficiaries of such a scheme
* Refusal of blood test
* Pregnant women

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiota assessment | 9 months
  At the end of the study, the analysis will be performed on all the samples at the same time by 16S RNAr pyrosequencing.

SECONDARY OUTCOMES:
Measuring the severity of ASD | 24 months
  The severity of ASD is evaluated by the ADOS2-CSS (Autism Diagnostic Observation Schedule-Calibrated Standardized Score) scale. A ADOS-CSS 4 score indicates a light TSA. It is moderate if the ADOS-CSS is between 5 and 7, and severe if it is greater than or equal to 8.
Evaluation of the level of social interaction | 24 months
  This level is evaluated by the parental questionnaire SRS-2 (Social Responsiveness Scale-2). This scale consists of 65 items. Each item is rated from 0 (never) to 3 (almost always true).
Behavioural disorders | 24 months
  These disorders are evaluated by the parental questionnaire ABC (Aberrant Behavior Checklist). This scale consists of 58 items. Items are rated from 0 (no problem) to 3 (severe problem).
Quality of life of children with ASD | 24 months
  The quality of life is evaluated by the parental questionnaire Kidscreen-27. This parental questionnaire consists of 27 items. Each item is rated from 0 to 4 (not always, to very often).
Developmental trajectory of children with ASD | 24 months
  This is evaluated by the scale Vineland II. The Vineland Scale is a 30-minute to an hour semi-structured interview administered with the child's parents. This scale is used to measure the subject's socio-adaptive abilities. Standard scores are obtained in three areas: communication, life skills and socialization. it consists of 577 items.
IQ (Intellectual Quotient) | 24 months
  This is evaluated by psychometric tests adapted to the children.
Assessment of stools aspect | 24 months
  This is assessed by Bristol stool scale. There is 7 types of stools to classify the consistency. The Bristol scale is a visual scale for classifying human stool according to its consistency, which depends on the time spent in the colon.
Repetitive and stereotypical behaviours | 24 months
  These behaviors are evaluated by the parental questionnaire RBS-R (Repetitive Behavior Scale reviewed)
Intensity of GI disorders | 24 months
  This is assessed by parental questionnaire PedsQL GSS (Gastrointestinal Symptom Scale)
Measurement of neuroinflammation | 9 months
  Measurement of neuroinflammation by serum immunological assays of a panel of 37 neuroinflammation markers (ELISA) consisting of cytokines, chemokines, markers of inflammation, angiogenesis and vascular lesion
Intestinal permeability | 9 months
  This is assessed by plasma assays of the following markers: zonulin and citrulline
Intestinal inflammation | 9 months
  This is assessed by plasma assays of marker I-FABP
Intestinal inflammation | 9 months
  This is assessed by plasma assays of marker LBP
Intestinal inflammation | 9 months
  This is assessed by plasma assays of marker sCD14
TH1/TH2 immune response | 9 months
  It will be done by assaying the different immune cell lines
Metabolome analysis | 9 months
  Assessment of nutritional status by Simultaneous quantification of routinely measured lipids as well as 14 categories of lipoproteins, fatty acid composition, glycolysis precursors, ketones, and amino acids will be performed using a suitable metabolomic NMR platform.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie MIOT, MD-PH, Principal Investigator — Montpellier University Hospital
Locations (1):
- Centre de Ressources Autisme, Montpellier, France